CLINICAL TRIAL: NCT06766513
Title: Characterization of the Sleep-Wake Cycle in Traumatic Brain Injury Patients with a Disorder of Consciousness
Acronym: SLEEPDOC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL24_0936; 2024-A02567-40 (Other: ID-RCB)
Record Dates: First submitted 2024-12-16; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Trauma, Nervous System; Brain Trauma
Keywords: Traumatic brain injury; Disorders of consciousness; Vegetative State; Minimally Conscious State
MeSH Terms: conditions — Trauma, Nervous System; Brain Injuries, Traumatic; Consciousness Disorders; Persistent Vegetative State | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients in a vegetative state (Experimental)
  Interventions: Other: Actimetry; Other: Subjective assessments; Other: questionnaire
- Patients in a minimally conscious state (Experimental)
  Interventions: Other: Actimetry; Other: Subjective assessments; Other: questionnaire

INTERVENTIONS:
Other: Actimetry — actimetry will be performed continuously during these 104 hours.
Other: Subjective assessments — The subjective assessments of the patient's awake/sleep state will be collected every 2 hours during the night and at least 3 times during the day, for a total of at least 8 assessments per 24-hour period, over a duration of 104 consecutive hours (slightly more than 4 days, starting at midnight and ending at 8 :00 AM, to cover 4 full days and 4 full nights).
Other: questionnaire — MOCA : Montreal Cognitive Assessment
Other: questionnaire — SF-36 The Short Form (36)
Other: questionnaire — CRS-R (Coma Recovery Scale-Revised)
Other: questionnaire — GOSE (Glasgow Outcome Scale-Extended)
Other: questionnaire — GCS (Glasgow Coma Scale)

SUMMARY:
Each year in France, 160,000 peoples suffer from a mild or severe traumatic brain injury (TBI). Sleep plays a crucial role in the process of brain plasticity, which is essential for neurological and cognitive recovery. However, the sleep-wake cycle is rarely, if ever, evaluated in patients with TBI and consciousness disorders within Post-Resuscitation Rehabilitation Units (SRPR). Caregivers develop, on a daily basis, an intuitive understanding of the patient's overall condition. This expertise deserves to be validated using objective sleep assessment tools (actigraphy). If proven accurate, it could lead to the implementation of a sleep-wake cycle evaluation protocol within SRPRs.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Post-Resuscitation Rehabilitation Unit or the Neurological Intensive Care Unit
* Consciousness disorders: Vegetative State or Minimally Conscious State (according to the CRS-R)
* Traumatic brain injury
* Patient aged 18 years or older
* Presence of relatives able to express non-opposition to the study
* Subjects affiliated with a social security scheme (or beneficiaries)

Exclusion Criteria:

* Admission for status epilepticus
* Individuals admitted to a healthcare or social care facility for purposes other than research
* Adults under legal protection measures (guardianship, conservatorship)
* Individuals not affiliated with a social security scheme or not benefiting from a similar scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Subjective assessments | during 104 consecutive hours after enrollment
Actimetry | during 104 consecutive hours after enrollment

SECONDARY OUTCOMES:
Coma Recovery Scale-Revised | once a day for 6 to 5 days
Coma Recovery Scale-Revised | 3 months after the start of study
Coma Recovery Scale-Revised | 6 months after the start of study
Glasgow Coma Scale assessment | once a day for 6 to 5 days
Glasgow Coma Scale assessment | 3 months after the start of study
Glasgow Coma Scale assessment | 6 months after the start of study
Glasgow Outcome Scale-Extended assessment | 6 months after the start of study
Glasgow Outcome Scale-Extended assessment | 3 months after the start of study
Montreal Cognitive Assessment | 3 months after the start of study
Montreal Cognitive Assessment | 6 months after the start of study
Short Form 36 assessment | 3 months after the start of the study
Short Form 36 assessment | 6 months after the start of study

CONTACTS AND LOCATIONS:
Overall Officials: Jacques LUAUTE, Professor, Principal Investigator — Hôpital Neurologique Pierre Wertheimer, Service de Service de Rééducation Post-Réanimation; Florent GOBERT, Doctor, Principal Investigator — Hôpital Neurologique Pierre Wertheimer, Service de Réanimation Polyvalente Neurologique
Locations (1):
- Hôpital Neurologique Pierre Wertheimer, Service de Réanimation Polyvalente Neurologique, Bron, France, France

IPD SHARING:
Plan to Share IPD: Undecided